CLINICAL TRIAL: NCT06395090
Title: LIGHTBEAM-U01 Substudy 01B: A Phase 1/2 Substudy to Evaluate the Safety and Efficacy of Pembrolizumab in Combination With Investigational Agents in Pediatric and Young Adult Participants With Hematologic Malignancies or Solid Tumors
Brief Title: A Study of Pembrolizumab in Combination With Investigational Agents in Pediatric and Young Adult Participants With Hematologic Malignancies or Solid Tumors (MK-9999-01B/LIGHTBEAM-U01)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: development program discontinuation
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9999-01B; MK-9999-01B (Other: MSD); LIGHTBEAM-U01 (Other: MSD); 2023-507179-23 (Registry Identifier: EU CT); U1111-1295-3472 (Registry Identifier: UTN)
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Favezelimab + Pembrolizumab (Experimental): Participants will receive pembrolizumab and favezelimab via an intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 cycles. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Biological: Favezelimab
- Favezelimab/Pembrolizumab (Experimental): Participants will receive coformulated favezelimab/pembrolizumab via an IV infusion Q3W for up to 35 cycles. Each cycle is 21 days.
  Interventions: Biological: Favezelimab/Pembrolizumab
- Pembrolizumab + Vibostolimab (Experimental): Participants will receive pembrolizumab and vibostolimab via an IV infusion Q3W for up to 35 cycles. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Biological: Vibostolimab
- Pembrolizumab/Vibostolimab (Experimental): Participants will receive coformulated pembrolizumab/vibostolimab via an IV infusion Q3W for up to 35 cycles. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab/Vibostolimab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475
  Arms: Favezelimab + Pembrolizumab; Pembrolizumab + Vibostolimab
Biological: Favezelimab — IV infusion
  Arms: Favezelimab + Pembrolizumab
Biological: Favezelimab/Pembrolizumab — IV infusion
  Other Names: MK-4280A
  Arms: Favezelimab/Pembrolizumab
Biological: Vibostolimab — IV infusion
  Arms: Pembrolizumab + Vibostolimab
Biological: Pembrolizumab/Vibostolimab — IV infusion
  Other Names: MK-7684A
  Arms: Pembrolizumab/Vibostolimab

SUMMARY:
This study is a rolling arm study of pembrolizumab in combination with investigational agents in pediatric participants with relapsed or refractory classical Hodgkin lymphoma (cHL) solid tumors with microsatellite instability-high (MSI-H)/mismatch repair deficient (dMMR) or tumor mutational burden-high (TMB-H). This study will have 2 parts: a safety lead-in to demonstrate a tolerable safety profile and confirm a preliminary recommended phase 2 dose (RP2D) (Part 1) followed by an efficacy evaluation (Part 2). Participants will be assigned to a treatment arm (either Part 1 or Part 2) that is open for enrollment.

There will be no hypothesis testing in this study.

DETAILED DESCRIPTION:
The master screening protocol is MK-9999-U01.

ELIGIBILITY:
Inclusion Criteria:

* Must have 1 of the following histologically or cytologically confirmed diagnosis of Relapsed or refractory classical Hodgkin lymphoma (cHL) solid tumors that are microsatellite instability-high (MSI-H)/mismatch repair deficient (dMMR), or solid tumors that are tumor mutational burden-high (TMB-H)
* Must have recovered from all AEs from previous anticancer therapies
* Human immunodeficiency virus (HIV)-infected participants have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Received prior anticancer therapy with an anti-PD-1, anti-programmed cell death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (anti-PD-L2) in combination with either an Anti- lymphocyte-activation gene 3 (LAG-3) agent or an Anti- T-cell immunoreceptor with immunoglobulin (Ig) and ITIM domains (TIGIT) agent
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Known additional malignancy that is progressing or has required active treatment within the past 1 year
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Active infection requiring systemic therapy
* Concurrent active Hepatitis B and Hepatitis C virus infection
* History of allogenic tissue/solid organ transplant
* Has symptoms of or is being treated for graft versus host disease (GVHD)
* Has not adequately recovered from major surgery or have ongoing surgical complications
* Known tumors involving the brainstem

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Who Experience Dose-limiting Toxicities (DLTs) | Up to 21 days
  The number of participants who experience toxicities that are possibly, probably, or definitely related to study therapy; that meet pre-defined severity criteria; and result in a change in the given dose will be reported.
Parts 1 and 2: Number of Participants Who Report at Least 1 Adverse Event (AE) | Up to approximately 27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Parts 1 and 2 : Number of Participants Who Discontinue Study Drug Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Part 1: Area Under the Curve (AUC) | Cycle 1: Predose, postdose, 3, 8, and 15 days postdose; Cycle 2: predose; Cycle 4: predose and postdose; Cycle 5 predose; once predose every 4 cycles from Cycle 6 up to Cycle 35. A cycle is 21 days
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 1: Maximum Concentration (Cmax) | Cycle 1: Predose, postdose, 3, 8, and 15 days postdose; Cycle 2: predose; Cycle 4: predose and postdose; Cycle 5 predose; once predose every 4 cycles from Cycle 6 up to Cycle 35. A cycle is 21 days
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 1: Concentration in the Blood Immediately Before the Next Dose (Ctrough) | Cycle 1: Predose, postdose, 3, 8, and 15 days postdose; Cycle 2: predose; Cycle 4: predose and postdose; Cycle 5 predose; once predose every 4 cycles from Cycle 6 up to Cycle 35. A cycle is 21 days
  Blood samples will be collected at specified intervals for the determination of Ctrough.
Parts 1 and 2: Objective Response Rate (ORR) per Lugano Response Criteria by Blinded Independent Central Review (BICR) | Up to approximately 57 months
  ORR is defined as the percentage of participants who have a complete response (CR) or partial response (PR) and will be evaluated using computed tomography (CT) and positron emission tomography (PET)-CT. Response was assessed based on the International Working Group Criteria: Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters (SPD) for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Parts 1 and 2: ORR per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Investigator | Up to approximately 57 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by the investigator will be presented.

SECONDARY OUTCOMES:
Parts 1 and 2: ORR per Lugano Response Criteria by Investigator | Up to approximately 57 months
  DCR is defined as the percentage of the participants who have stable disease (SD), CR or PR. Response is assessed by CT and PET-CT and evaluated based on Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in SPD for up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% beyond normal). SD is no significant change from baseline in response and no criteria met for progressive disease. DCR as assessed by the investigator will be presented.
Parts 1 and 2: Disease Control Rate (DCR) per Lugano Response Criteria by BICR | Up to approximately 57 months
  DCR is defined, per RECIST 1.1, as the percentage of participants who have a CR: Disappearance of all target lesions or PR: At least a 30% decrease in the sum of diameters of target lesions or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.] The DCR as assessed by BICR will be presented.
Parts 1 and 2: DCR per RECIST 1.1 by Investigator | Up to approximately 57 months
  DCR is defined, per RECIST 1.1, as the percentage of participants who have a CR: Disappearance of all target lesions or PR: At least a 30% decrease in the sum of diameters of target lesions or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.] The DCR as assessed by BICR will be presented.
Parts 1 and 2: Duration of Response (DOR) per Lugano Response Criteria by BICR | Up to approximately 57 months
  For participants who demonstrate a confirmed CR or PR, DOR is defined as the time from CR or PR to documented disease progression or death. Participants are assessed using CT and PET-CT and response was evaluated based on the Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in SPD for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). DOR as assessed by BICR will be presented.
Parts 1 and 2: DOR per RECIST 1.1 by Investigator | Up to approximately 57 months
  For participants who demonstrate a confirmed CR: disappearance of all target lesions or PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by the investigator will be presented.
Parts 1 and 2: Progression Free Survival (PFS) per Lugano Response Criteria by BICR | Up to approximately 57 months
  PFS is defined as the time from randomization to documented disease progression or death, whichever occurs first as based on Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). PFS as assessed by BICR will be presented.
Parts 1 and 2: PFS per RECIST 1.1 by Investigator | Up to approximately 57 months
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by the investigator will be presented.
Parts 1 and 2: Overall Survival (OS) | Up to approximately 57 months
  OS is defined as time from first dose of study treatment to death due to any cause.
Part 2: Area Under the Curve (AUC) | Cycle 1: Predose, postdose, 3, 8, and 15 days postdose; Cycle 2: predose; Cycle 4: predose and postdose; Cycle 5 predose; once predose every 4 cycles from Cycle 6 up to Cycle 35. A cycle is 21 days
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 2: Maximum Concentration (Cmax) | Cycle 1: Predose, postdose, 3, 8, and 15 days postdose; Cycle 2: predose; Cycle 4: predose and postdose; Cycle 5 predose; once predose every 4 cycles from Cycle 6 up to Cycle 35. A cycle is 21 days
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 2: Concentration in the Blood Immediately Before the Next Dose (Ctrough) | Cycle 1: Predose, postdose, 3, 8, and 15 days postdose; Cycle 2: predose; Cycle 4: predose and postdose; Cycle 5 predose; once predose every 4 cycles from Cycle 6 up to Cycle 35. A cycle is 21 days
  Blood samples will be collected at specified intervals for the determination of Ctrough.
Parts 1 and 2: Antidrug Antibody (ADA) Levels | Cycle 1, 2, 4, and 5: predose; once every four cycles from Cycle 6 up to Cycle 35. A cycle is 21 days
  Blood samples will be collected at specified intervals for the determination of ADA levels.
Parts 1 and 2: Biomarker Levels for Classical Hodgkin Lymphoma (cHL) | Up to approximately 57 months
  For participants with cHL, the biomarker levels for cHL will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (12):
- United States (9):
  - Yale-New Haven Hospital ( Site 2012), New Haven, Connecticut
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 2017), Iowa City, Iowa
  - Children's Mercy Hospital ( Site 2024), Kansas City, Missouri
  - Rutgers Cancer Institute of New Jersey ( Site 2008), New Brunswick, New Jersey
  - New York Medical College ( Site 2023), Valhalla, New York
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 2003), Fargo, North Dakota
  - Children's Hospital of Philadelphia (CHOP) ( Site 2021), Philadelphia, Pennsylvania
  - Sanford Children's Hospital-Sanford Children's Specialty Clinic ( Site 2015), Sioux Falls, South Dakota
  - Intermountain - Primary Children's Hospital ( Site 2014), Salt Lake City, Utah
- South Korea (2):
  - Seoul National University Hospital-Pediatrics ( Site 2972), Seoul
  - Asan Medical Center-Pediatrics - Pedicatric Oncology ( Site 2973), Seoul
- National Taiwan University Hospital ( Site 2983), Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26121&tenant=MT_MSD_9011